CLINICAL TRIAL: NCT07147400
Title: Phase 2 Randomized, Double-blind, Controlled Study of Pfs230D1-CRM197 With R21 in Matrix-M1 in Healthy African School Children and Adults
Brief Title: Pfs230D1 + R21 in Matrix-M1 in African School Children and Adults
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Serum Institute of India Pvt. Ltd. (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VIMT 002
Record Dates: First submitted 2025-08-12; First posted 2025-08-29 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Prevention of Malaria Transmission and Clinical Malaria
MeSH Terms: interventions — Matrix-M; Adjuvants, Pharmaceutic

STUDY DESIGN:
Intervention Model Description: 1200 Healthy male and non-pregnant female participants of age 9-50 years will be enrolled in VIMT002 study in Bancoumana, Mali and surrounding villages.
  Participants aged 9 - 17 years in the immunobridging cohort (n=540) will be randomized to one of the study arms (2:2:1:1) to receive 10µg R21 in 50µg of Matrix-M1 single vial formulation, control vaccine (RABIVAX-S), or 6µg Pfs230D1-CRM197 with 10µg R21 in 50µg of Matrix-M1 as either a bedside mixture or a single-vial coformulation.
  Participants in the main cohort will be randomized to one of the study arms (1:1:1) to receive 10µg R21 in 50µg of Matrix-M1, control vaccine (RABIVAX-S), or 6µg Pfs230D1-CRM197 with 10 µg R21 in 50µg of Matrix-M1 single-vial coformulation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be conducted with a double blind. Because there is some variation in vaccine volumes, the unblinded pharmacy team will cover all syringes (after vaccine preparation) with opaque tape to maintain blinding. The participants, the clinical staff, laboratory staff and the study team involved in study endpoint assessments will be blinded to study treatment allocation. An additional layer to be implemented to promote blinding is that designated clinical staff who administer the vaccinations will only participate in study product administration and will remain separate from the team of blinded investigators who conduct all subsequent follow-up study assessments. The pharmacy team at the study site where vaccine preparation and administration is taking place will be unblinded, and they are responsible for maintaining security of study treatment assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Arm 1a (n=180), 9-17 years of age, Immunobridging cohort (Experimental): 10µg of R21 with 50µg Matrix-M1
  Interventions: Biological: 10µg of R21 with 50µg Matrix-M1
- Arm 2a (n=180), 9-17 years of age, Immunobridging cohort (Experimental): Control vaccine (rabies vaccine)
  Interventions: Biological: RABIVAX-S
- Arm 3a (n=90), 9-17 years of age, Immunobridging cohort (Experimental): 6µg of Pfs230D1-CRM197 + 10µg of R21 with 50µg Matrix-M1 single vial coformulation
  Interventions: Biological: 6µg of Pfs230D1-CRM197 + 10µg of R21 with 50µg Matrix-M1 single vial coformulation
- Arm 4a (n=90), 9-17 years of age, Immunobridging cohort (Experimental): 6µg of Pfs230D1-CRM197 + 10µg of R21 with 50µg Matrix-M1 bedside mix
  Interventions: Biological: Conjugated Pfs230D1 Vaccine (Pfs230D1-CRM197) For Bedside Mixing; Biological: R21 Malaria Vaccine (Recombinant) For Bedside Mixing; Biological: MATRIX-M1 (Adjuvant) For Bedside Mixing
- Arm 1b (n=120), 9-17 years of age, main cohort (Experimental): 10µg of R21 with 50µg Matrix-M1
  Interventions: Biological: 10µg of R21 with 50µg Matrix-M1
- Arm 2b (n=120), 9-17 years of age, main cohort (Experimental): Control vaccine (rabies vaccine)
  Interventions: Biological: RABIVAX-S
- Arm 3b (n=120), 9-17 years of age, main cohort (Experimental): 6µg of Pfs230D1-CRM197 + 10µg of R21 with 50µg Matrix-M1 single vial coformulation
  Interventions: Biological: 6µg of Pfs230D1-CRM197 + 10µg of R21 with 50µg Matrix-M1 single vial coformulation
- Arm 1c (n=100), 18-50 years of age, main cohort (Experimental): 10µg of R21 with 50µg Matrix-M1
  Interventions: Biological: 10µg of R21 with 50µg Matrix-M1
- Arm 2c (n=100), 18-50 years of age, main cohort (Experimental): Control vaccine (rabies vaccine)
  Interventions: Biological: RABIVAX-S
- Arm 3c (n=100), 18-50 years of age, main cohort (Experimental): 6µg of Pfs230D1-CRM197 + 10µg of R21 with 50µg Matrix-M1 single vial coformulation
  Interventions: Biological: 6µg of Pfs230D1-CRM197 + 10µg of R21 with 50µg Matrix-M1 single vial coformulation

INTERVENTIONS:
Biological: 10µg of R21 with 50µg Matrix-M1 — R21 is a portion of Pf circumsporozoite protein fused with hepatitis B surface antigen in the form of non-infectious virus-like particles (VLPs) produced in yeast cells (Hansenula) by recombinant DNA technology. Matrix-M1 (Adjuvanted) is cGMP manufactured by Serum Institute of India, PVD, LTD (SIIPL), Pune.
  Arms: Arm 1a (n=180), 9-17 years of age, Immunobridging cohort; Arm 1b (n=120), 9-17 years of age, main cohort; Arm 1c (n=100), 18-50 years of age, main cohort
Biological: 6µg of Pfs230D1-CRM197 + 10µg of R21 with 50µg Matrix-M1 single vial coformulation — R21 Malaria antigen is expressed in a recombinant high expressing Hansenula polymorpha production strain. The R21 Malaria drug substance lots/batches were cGMP manufactured at SIIPL, India.
  Recombinant CRM197 is a recombinant protein, and its drug substance lots/batches cGMP manufactured using Pseudomonas fluorescens production strain at SIIPL, India.
  Recombinant Pfs230D1M drug substance lots/batches of cGMP were manufactured using Hansenula Polymorpha and manufactured at the SIIPL.
  A single vial coformulation containing 10µg R21 and 6µg Pfs230D1-CRM197 conjugate mixed with 50µg Matrix-M1 has been developed and is manufactured by SIIPL.
  Arms: Arm 3a (n=90), 9-17 years of age, Immunobridging cohort; Arm 3b (n=120), 9-17 years of age, main cohort; Arm 3c (n=100), 18-50 years of age, main cohort
Biological: RABIVAX-S — Sterile, purified inactivated rabies vaccine prepared on vero cells, indicated for the prevention of rabies in children and adults.
  Arms: Arm 2a (n=180), 9-17 years of age, Immunobridging cohort; Arm 2b (n=120), 9-17 years of age, main cohort; Arm 2c (n=100), 18-50 years of age, main cohort
Biological: Conjugated Pfs230D1 Vaccine (Pfs230D1-CRM197) For Bedside Mixing — Recombinant Pfs230D1M drug substance lots/batches cGMP manufactured using Pichia pastoris manufactured at the Pilot Bioproduction Facility, Walter Reed Army Institute of Research (Silver Spring, Maryland), and at SIIPL respectively.
  Recombinant CRM197 is a recombinant protein and its drug substance lots/batches cGMP manufactured using Pseudomonas fluorescens production strain at SIIPL, India.
  Arms: Arm 4a (n=90), 9-17 years of age, Immunobridging cohort
Biological: R21 Malaria Vaccine (Recombinant) For Bedside Mixing — R21 is a fusion protein of hepatitis B surface antigen (HBsAg) to the C-terminus and central repeats of the circumsporozoite (CS) protein of Plasmodium falciparum. R21 VLP, recombinant HBsAg spontaneously self-assembled & formed a virus-like particle, wherein circumsporozoite protein (CSP) from Plasmodium falciparum is presented on the VLP of recombinant HBsAg particles. R21 Malaria antigen expressed in recombinant high expressing Hansenula polymorpha production strain. The R21 Malaria drug substance lots/batches were cGMP manufactured at SIIPL, India.
  Arms: Arm 4a (n=90), 9-17 years of age, Immunobridging cohort
Biological: MATRIX-M1 (Adjuvant) For Bedside Mixing — active ingredient in Matrix-M1 are saponin-based fractions. Matrix-M1 has a ratio of Matrix-A and Matrix-C of 85:15 (by weight). Both Matrix-A and Matrix-C are individual fractions (separated by chromatography) derived from extracts from the Quillaja saponaria tree. Matrix-M1 (Adjuvanted) is cGMP manufactured by Serum Institute of India, PVD, LTD (SIIPL), Pune.
  Arms: Arm 4a (n=90), 9-17 years of age, Immunobridging cohort

SUMMARY:
This is a Phase 2, randomized, double-blind, controlled study designed to evaluate the safety, tolerability, immunogenicity, vaccine efficacy, and functional activity of Pfs230D1-CRM197 conjugate vaccine with R21 nanoparticle vaccine formulated on Matrix-M1. Participants (9-50 years of age) will be drawn from Bancoumana, Mali and the surrounding areas.

DETAILED DESCRIPTION:
Participants aged 9 - 17 years in the immunobridging cohort (n=540) will be randomized to one of the study arms ( 2:2:1:1) to receive 10μg R21 alone in 50μg of Matrix-M1, control vaccine (RABIVAX-S), or 6μg Pfs230D1-CRM197 with 10μg R21 in 50μg of Matrix-M1 as either a bedside mixture or a single-vial coformulation.

Participants in the main cohort who are aged 9-17 years will be randomized to one of the study arms (1:1:1) to receive 10μg R21 alone in 50μg of Matrix-M1, control vaccine (RABIVAX-S), or 6μg Pfs230D1-CRM197 with 10 μg R21 in 50μg of Matrix-M1 single-vial coformulation. Enrollment of participants aged 9-17 years in the main cohort will be done after DSMB reviews the 7-day safety data post dose 1 from the immunobridging cohort.

Participants in the main cohort who are aged 18 - 50 years will be randomized to one of the study arms (1:1:1) to receive either 10μg R21 alone in 50μg of Matrix-M1, control vaccine (RABIVAX-S), or 6μg Pfs230D1-CRM197 with 10μg R21 in 50μg of Matrix-M1 single-vial coformulation.

Enrollment of adult participants aged 18 -50 years in the main cohort (n=300) will be done from the start of the study and will be independent of enrollment into of the pediatric cohort (9-17 years).

All vaccines will be administered as an intramuscular (IM) injection on a 0, 28, 56 day schedule with an option for additional follow-up for a subsequent malaria transmission season with or without a fourth dose approximately 52 weeks after the third vaccine dose (based on year 1 results).

Initial enrollment will be staggered over time for safety, but all participants will be analyzed together for primary, secondary, and exploratory endpoints.

A total 1200 participants will be randomized into the study as below:

Immunobridging cohort (Participants 9-17 years of age, n = 540) (2:2:1:1 randomization)

* Arm 1a (n = 180): 10µg of R21 with 50µg Matrix-M1 on study day 0, 28, 56 +/- 392
* Arm 2a (n = 180): Control vaccine (rabies vaccine) on study day 0, 28, 56 +/- 392
* Arm 3a (n = 90): 6µg of Pfs230D1-CRM197 + 10µg of R21 with 50µg Matrix-M1 single vial coformulation on study day 0, 28, 56 +/- 392
* Arm 4a (n = 90): 6µg of Pfs230D1-CRM197 + 10µg of R21 with 50µg Matrix-M1 bedside mix on study day 0, 28, 56 +/- 392

Main cohort:

Participants 9-17 years of age (n = 360) (1:1:1 randomization):

* Arm 1b (n=120): 10µg of R21 with 50µg Matrix-M1 on study day 0, 28, 56 +/- 392
* Arm 2b (n = 120): Control vaccine (rabies vaccine) on study day 0, 28, 56 +/- 392
* Arm 3b (n = 120): 6µg of Pfs230D1-CRM197 + 10µg of R21 with 50µg Matrix-M1 single vial coformulation on study day 0, 28, 56 +/- 392

Participants 18-50 years of age (n = 300) (1:1:1 randomization):

* Arm 1c (n=100): 10µg of R21 with 50µg Matrix-M1 on study day 0, 28, 56 +/- 392
* Arm 2c (n = 100): Control vaccine (rabies vaccine) on study day 0, 28, 56 +/- 392
* Arm 3c (n = 100): 6µg of Pfs230D1-CRM197 + 10µg of R21 with 50µg Matrix-M1 single vial coformulation on study day 0, 28, 56 +/- 392

ELIGIBILITY:
Inclusion Criteria:

1. Age:>/= 9 years old and </= 50 years old.
2. Provides written informed consent if >/=18 years of age.
3. Provides written informed consent of parent/guardian if <18 years of age, with additional participant written assent obtained from children > 12 years of age.
4. Known resident or long-term resident (more than 1 year) of trial site or surrounding villages.
5. Available for the duration of the trial.
6. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
7. In good general health and without clinically significant medical history in the opinion of the investigator.
8. Permission for long term storage of blood samples.

   • Note: If a participant withdraws consent or at the time of study completion or end of participation wishes to withdraw permission for long term storage of blood samples, this can be requested, and sample destruction will be documented.
9. Females of reproductive potential aged 12 years and above who have attained menarche and are sexually active must be willing to use reliable contraception from 21 days prior to Study Day 1 and 21 days prior to Study Day 392 (booster dose) and until 1 month after the last vaccination in primary series and after booster dose.

   * A reliable method of birth control includes one of the following:

     * Confirmed pharmacologic contraceptives (parenteral) delivery.
     * Intrauterine or implantable device.
     * Barrier methods.

EXCLUSION CRITERIA:

1. Pregnant and breastfeeding females. Pregnant, as determined by a positive urine or serum beta human choriogonadotropin (βhCG) test.

   NOTE: Pregnancy is also a criterion for discontinuation of any further vaccine dosing
2. Menstruating females less than 12 years of age. (In order to avoid cultural implications of further assessing pregnancy potential i.e. sexual activity in this age group).

   NOTE: If a female less than 12 years of age starts menarche while on study it will not be exclusionary for them to continue participation, but will undergo pregnancy testing prior to each vaccination.
3. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and comply with the study protocol at a level appropriate for the participant's age.
4. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies including urinalysis.
5. Current or planned participation in an investigational product study until the time period of the last required study visit under this protocol.
6. Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
7. History of a severe allergic reaction or anaphylaxis.
8. Known:

   * Severe asthma, defined as asthma that is unstable or required emergent care, urgent care, hospitalization, or intubation during the past 2 years, or that has required the use of oral or parenteral corticosteroids at any time during the past 2 years.
   * Autoimmune or antibody-mediated disease including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjögren's syndrome, or autoimmune thrombocytopenia.
   * Immunodeficiency.
   * Seizure disorder (exception: history of simple febrile seizures).
   * Asplenia or functional asplenia.
   * Use of chronic (≥14 days) oral or intravenous (IV) corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone >10 mg/day) or immunosuppressive drugs within 30 days of enrollment.
   * Hypersensitivity reaction to rabies vaccine in the past.
9. Receipt of:

   * Live vaccine within 4 weeks prior to enrollment or a killed vaccine within 2 weeks prior to enrollment.
   * Immunoglobulins and/or blood products within the past 3 months.
   * Any malaria vaccine in the past.
   * Any investigational product in the last 6 months
10. Any other condition that in the opinion of the investigator might jeopardize the safety or rights of a participant participating in the trial, interfere with the evaluation of the study objectives, or might render the participant unable to comply with the protocol.

Ages: 9 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Immediate adverse events in all participants | Up to 30-minutes following each dose
  Occurrence of immediate adverse events
Number of Participants with solicited local adverse events in reactogenicity group | Up to 7 days following each dose
  Occurrence of solicited local adverse events
Number of Participants with Solicited systemic adverse events in reactogenicity group | Up to 7 days following each dose
  Occurrence of solicited systemic adverse events
Number of Participants with Unsolicited adverse events in all participants | Up to 28 days following each vaccination
  Occurrence of unsolicited adverse events
Number of Participants with Serious adverse events in all participants | Through the whole study duration, 24 months post dose 3 or 12 months post dose 4
  Occurrence of serious adverse events
Number of Participants with Abnormal Laboratory Values post-vaccination in laboratory safety group | at 7 days following each vaccination
  Laboratory adverse events
Anti-NANP IgG antibodies | at 4 weeks post dose 3
  Antibody responses to NANP IgG antibodies
Anti-Pfs230D1 IgG antibodies | at 4 weeks post dose 3
  Antibody responses to Pfs230D1 IgG antibodies

SECONDARY OUTCOMES:
To assess vaccine functional activity against transmission by DSF | from 2 weeks to 24 weeks after completion of the primary vaccine course +/- booster
  Proportion reduction in proportion of infected mosquitoes (among those dissected)
To assess vaccine functional activity against transmission by DSF | from 2 weeks to 24 weeks after completion of the primary vaccine course +/- booster
  Proportion reduction in DSFs with at least one infected mosquito
humoral immunogenicity time trends and durability | at baseline, 28 days after each dose and through study completion, at an average of 1 month
  Antibody responses to Pfs230D1
humoral immunogenicity time trends and durability | at baseline, 28 days after each dose and through study completion, at an average of 1 month
  Antibody responses to NANP
To assess the protective efficacy against clinical malaria caused by Pf | At 24 and 52 weeks after completion of the primary and booster vaccine course
  Efficacy against clinical malaria as defined by: presence of asexual P. falciparum parasitemia >0 parasites/µL and/or RDT positive with either an axillary temperature of ≥37.5 °C or one or more of the following symptoms: history of fever within the last 48 hours, headache, myalgia, arthralgia, malaise, nausea, dizziness, or abdominal pain

CONTACTS AND LOCATIONS:
Locations (1):
- University of Science, Technique and Technology of Bamako (Usttb), Bamako, Mali

IPD SHARING:
Plan to Share IPD: No